CLINICAL TRIAL: NCT01257087
Title: Resolution of Type 2 Diabetes Mellitus: Intensive vs. Conventional Glycaemic Control After Obesity Surgery.
Acronym: GLUCOSURG1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Principal Investigator, Carel Le Roux, Consultant metabolic medicine, Imperial College London
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLUCOSURG1
Record Dates: First submitted 2010-12-08; First posted 2010-12-09 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-10

CONDITIONS: Type 2 Diabetes Mellitus; Obesity
Keywords: Type 2 Diabetes Mellitus; Obesity; Bariatric Surgery; Glycaemic control; Microvascular complications; Intensive; Conservative
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Insulin; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive glycaemic control (Experimental): Intensive glycaemic control All patients will be prescribed insulin glargine once a day. The dose of the insulin will be adjusted to achieve fasting capillary glucose levels between 5-7 in the intensive group and 7-9 mmol/l in the control group.
  Interventions: Drug: Insulin
- Conservative glycaemic control (Active Comparator): Conservative glycaemic control All patients will be prescribed insulin glargine once a day. The dose of the insulin will be adjusted to achieve fasting capillary glucose levels between 5-7 in the intensive group and 7-9 mmol/l in the control group.
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — All patients will be prescribed insulin glargine once a day. The dose of the insulin will be adjusted to achieve fasting capillary glucose levels between 5-7 in the intensive group and 7-9 mmol/l in the control group.
  Other Names: Insulin Glargine

SUMMARY:
Obesity surgery is very effective in improving or even curing Type 2 Diabetes in patients with obesity. Many patients stop or reduce their medication after surgery and this can happen fairly quickly. The investigators do not know whether strict control of blood glucose/sugar after the operation makes any difference in the long term. Additionally many patients prefer their blood sugars to be a "bit high" because they are afraid of hypos.A number of studies have described patients whose eye, nerve and kidney disease has deteriorated when high sugars are controlled very quickly. The investigators want to ensure that surgery provides maximum benefit and remains safe in patients with diabetes. This study will help us decide if the investigators should be strict with blood glucose after obesity surgery operations or not and whether obesity surgery is safe for the eye, nerve and kidney complications of diabetes.

DETAILED DESCRIPTION:
Subjects would be randomised into intensive glycaemic control and conventional glycaemic control after obesity surgery. Data on complications of diabetes such as eye, nerve and kidney will be collected before obesity surgery and 1 year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 2 Diabetes Mellitus who have been approved for obesity surgery

Exclusion Criteria:

* Patients with Type 2 Diabetes Mellitus who do not require insulin immediately after obesity surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-12; Primary Completion 2016-02 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carel W le Roux, MRCP, PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intensive Glycaemic Control | Conservative Glycaemic Control
Started | 18 | 17
Completed | 18 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Not differenet
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensive Glycaemic Control | Conservative Glycaemic Control | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 55 (6) | 49 (7) | 52 (6.5)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 5 | 10 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 18 | 17 | 35
  Unknown or Not Reported | 0 | 0 | 0
HbA1C [Mean (Standard Deviation); unit: %] | 8.7 (1.2) | 8.8 (1.0) | 8.75 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Type 2 Diabetes Mellitus Who Achieve Fasting Blood Glucose of Less Than 5.6 mmol/l and/or HbA1c of Less Than 6%
Description: Patients will be tested off all anti-diabetes medications if safe to do so to assess the percentage of patients with Type 2 Diabetes Mellitus who achieve fasting blood glucose of less than 5.6 mmol/l and/or HbA1c of less than 6%
Time Frame: 1 year after surgery
Population: not different
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive Glycaemic Control | Conservative Glycaemic Control
Number analyzed (Participants) | 18 | 17
Participants | 4 | 4

2. Secondary Outcome: Percentage of Type 2 Diabetes Mellitus Patients With a Reduction in the Doses/Number of Diabetes Medications Used Preoperatively
Description: A list of patients medication will be collected to assess the percentage of Type 2 Diabetes Mellitus patients with a reduction in the doses/number of diabetes medications used preoperatively
Time Frame: 1 year after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive Glycaemic Control | Conservative Glycaemic Control
Number analyzed (Participants) | 18 | 17
Participants | 18 | 17

3. Secondary Outcome: Number of Participants With Microvascular Events
Description: Composite of microvascular events will be defined as new or worsening nephropathy, retinopathy or neuropathy.
Time Frame: 1 year after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive Glycaemic Control | Conservative Glycaemic Control
Number analyzed (Participants) | 18 | 17
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: Not different
Arm/Group | Intensive Glycaemic Control | Conservative Glycaemic Control
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 1/18 | 1/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intensive Glycaemic Control (N=18) | Conservative Glycaemic Control (N=17)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes